CLINICAL TRIAL: NCT01420172
Title: Pulmonary Disease in Patients Undergoing Hematopoietic Stem Cell Transplantation.
Status: Completed | Type: Observational
Sponsor: Karen Wood (Other)
Responsible Party: Sponsor-Investigator, Karen Wood, MD, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2011H0214
Record Dates: First submitted 2011-08-16; First posted 2011-08-19 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2015-10

CONDITIONS: Post Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post hematopoietic stem cell transplantation: Patients who were seen post hematopoietic stem cell transplantation between 01Jan2000 and 30Jun2011
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Collection of data on patients who were seen at OSUMC at any time between 01Jan2000 and 30Jun2011 post hematopoietic stem cell transplantation

SUMMARY:
This will be a retrospective study and analysis of subjects who have undergone a hematopoietic stem transplant (either at OSUMC or external location) and were seen at OSUMC at any time between 01Jan2000 and 30Jun2011.

This study will determine factors influencing pulmonary disease and associated treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have undergone a hematopoietic stem transplant (either at OSUMC or external location) and were seen at OSUMC at any time between 01Jan2000 and 30Jun2011.
* Age > 18 years

Exclusion Criteria:

* Age <18 years
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient record captured during 01Jan2000 and 30Jun2011 from the medical record at The Ohio State University Medical Center who were seen post hematopoietic stem transplant.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-08; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

PRIMARY OUTCOMES:
A retrospective diagnostic review on pulmonary disease related to hematopoietic stem cell transplantation. | Up to 15 years
  To determine factors influencing pulmonary disease related to HSCT.

SECONDARY OUTCOMES:
A retrospective treatment review on treatment strategies for pulmonary disease related to hematopoietic stem cell transplantation. | Up to 15 years
  To review treatment strategies for pulmonary disease post transplant for effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Afessa B, Litzow MR, Tefferi A. Bronchiolitis obliterans and other late onset non-infectious pulmonary complications in hematopoietic stem cell transplantation. Bone Marrow Transplant. 2001 Sep;28(5):425-34. doi: 10.1038/sj.bmt.1703142. PMID 11593314
- [Background] Williams KM, Chien JW, Gladwin MT, Pavletic SZ. Bronchiolitis obliterans after allogeneic hematopoietic stem cell transplantation. JAMA. 2009 Jul 15;302(3):306-14. doi: 10.1001/jama.2009.1018. PMID 19602690
- [Background] Dudek AZ, Mahaseth H, DeFor TE, Weisdorf DJ. Bronchiolitis obliterans in chronic graft-versus-host disease: analysis of risk factors and treatment outcomes. Biol Blood Marrow Transplant. 2003 Oct;9(10):657-66. doi: 10.1016/s1083-8791(03)00242-8. PMID 14569562
- [Background] Verleden GM, Vanaudenaerde BM, Dupont LJ, Van Raemdonck DE. Azithromycin reduces airway neutrophilia and interleukin-8 in patients with bronchiolitis obliterans syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):566-70. doi: 10.1164/rccm.200601-071OC. Epub 2006 Jun 1. PMID 16741151
- [Background] Vos R, Vanaudenaerde BM, Verleden SE, De Vleeschauwer SI, Willems-Widyastuti A, Van Raemdonck DE, Schoonis A, Nawrot TS, Dupont LJ, Verleden GM. A randomised controlled trial of azithromycin to prevent chronic rejection after lung transplantation. Eur Respir J. 2011 Jan;37(1):164-72. doi: 10.1183/09031936.00068310. Epub 2010 Jun 18. PMID 20562124